CLINICAL TRIAL: NCT03468491
Title: The Additional Effect of First Metatarsophalangeal Joint Correction on Runners With First Ray Instability and Patellofemoral Pain Syndrome
Brief Title: The Additional Effect of Hallux Valgus Correction on Runners With First Ray Instability and Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YM106048F
Record Dates: First submitted 2018-02-06; First posted 2018-03-16 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2018-05

CONDITIONS: Patellofemoral Pain Syndrome; Hallux Valgus
Keywords: Patellofemoral pain syndrome; Runner; First ray instability; Lower extremity closed chain exercise
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Hallux Valgus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined training group (Experimental): Biomechanical taping will first being applied to the participants of the combined training group. They will be asked to perform following exercises in this session afterwards. As the treatment session goes on, a set of foot intrinsic muscle strengthening exercise and lower extremity neuromuscular exercise will be provided.
  Interventions: Other: combined training
- Proximal training group (Active Comparator): For participants of the proximal training group, only a set of lower extremity neuromuscular exercise will be provided. This set of exercises is designed to be the same as for participants of combined training group.
  Interventions: Other: Proximal training

INTERVENTIONS:
Other: combined training — The whole intervention period will last for 6 weeks, 2 visits per week, 1 hour per visit in the Research Building Room 630 of National Yang Ming University. All programs will be under the supervision of a physiotherapist with 2-year experience individually. 1. Hallux valgus correction: 1.1 Joint alignment correction (Grade II joint mobilization, 10 times/set, 3 sets/visit) - 1st MTP joint distraction - Proximal talofibular joint anteroposterior glide - (Grade III joint mobilization if any restriction being found) 1.2 Biomechanical taping (using Dynamic taping, 1 time/ visit, keep the taping for 2 days minimum) 1.3 Foot intrinsic muscle strengthening (10 times/set for each exercise, 3 sets/visit): - Short foot exercise - Toespread out exercise - Heel-rise exercises 2. Lower extremity neuromuscular exercises: (10-15 times/set, 3 sets/visit) 2.1 Single lunge 2.2 Stepping down 2.3 Vertical squat 2.4 Vertical jumping
  Other Names: hallux valgus correction; lower extremity neuromuscular exercises
  Arms: Combined training group
Other: Proximal training — 1. Lower extremity neuromuscular exercises: (10-15 times/set, 3 sets/visit) 1.1 Single lunge 1.2 Stepping down 1.3 Vertical squat 1.4 Vertical jumping All exercises will first start on firm surface without additional resistance/weight. Later, settings will be gradually shifted into on firm surface with resisted band from random direction, on a cushion with/ without resisted band, on a BOSU balance trainer. Progression are made every 2 weeks ideally, while adjustments may be taken into concern due to individual differences.
  Other Names: lower extremity neuromuscular exercises
  Arms: Proximal training group

SUMMARY:
The study purpose is to investigate the effectiveness of a program combining biomechanical taping with lower extremity neuromuscular exercises for runners with patellofemoral pain syndrome (PFPS) and hallux valgus

DETAILED DESCRIPTION:
This will be a single-blind, experimental study with two treatment groups. A total of 30 college athletes with PFPS and hallux valgus and majoring in long distance running or soccer, or recreational runners in Taipei metropolitan area will be recruited. A set of clinical examination will be conducted to rule out abnormal knee structures, pathologies, or injuries apart from PFPS. The lower extremity alignment as well as hip and knee kinematics during a step down test will be tracked using Noraxon's myoMOTION system. Muscle activation of the muscles controlling the hip and knee movements during the step down test will be recorded using TELEmyo DTS of Noraxon. Hallux valgus angle will be measured with surface markers on photographs. Knee pain level will be rated in a visual analog scale. The investigators will analyze the data with Statistical Product and Service Solutions (SPSS) for Windows. Repeated-measure ANOVAs will be used to examine group-by-time interaction on all the outcome variables. All significance level will be set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* High physical activity level (running at least 5 times/week and at least 2 hours/time)
* Presenting anterior/retropatellar knee pain in the past 6 months
* At least two of the following activities provocated symptom: Prolonged sitting, ascending and/or descending stairs, squatting, kneeling, running, limping
* Not having any pathologies of knee joint (ligament tear, menisci injury, patellofemoral joint dislocation, tendinitis, bursitis…etc.)
* With hallux valgus angle>15°
* With 1st metatarsophalangeal joint instability
* 20~40 y/o

Exclusion Criteria:

* Lower extremities osteoarthritis
* Systematic diseases such as rheumatoid arthritis, systemic lupus erythematosus, DM…etc.
* Lower extremities fracture history
* Surgical history of lower extremities
* Neurological pathology that would interfere with gait
* Hallux could not be corrected to neutral through passive correction
* Low back pain and/or sacroiliac joint dysfunction in the past six months
* Excessive femoral anteversion

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Displacement of femur in step-down test | changes from baseline and after 6 weeks of intervention
  displacement recorded in cm/BMI
Displacement of tibia in step-down test | changes from baseline and after 6 weeks of intervention
  displacement recorded in cm/BMI
Knee pain level | changes from baseline and after 6 weeks of intervention
  The level of knee pain during daily activities will be quantified with visual analogue scale.
Changes of pain-free running distance | changes from baseline and after 6 weeks of intervention
  The changes of pain-free running distance will be recorded in kilometers.
EMG amplitude of knee extensor | changes from baseline and after 6 weeks of intervention
  amplitude recorded in %MVC
EMG amplitude of knee flexor | changes from baseline and after 6 weeks of intervention
  amplitude recorded in %MVC
EMG amplitude of hip external rotator | changes from baseline and after 6 weeks of intervention
  amplitude recorded in %MVC
changes of the muscle activation time between vastus medialis oblique and vastus lateralis | changes from baseline and after 6 weeks of intervention
  changes of the muscle activation time recorded in second

SECONDARY OUTCOMES:
Tibiofemoral angle in relaxed standing | changes from baseline and after 6 weeks of intervention
  recorded in degree
Hallux valgus angle in relaxed standing | changes from baseline and after 6 weeks of intervention
  recorded in degree
Navicular drop | changes from baseline and after 6 weeks of intervention
  navicular position changes between sitting and relaxed standing, recording in cm
Arch height index | changes from baseline and after 6 weeks of intervention
  arch height in one leg standing, recording in the ratio of arch height and truncated foot length
Hip rotation angle in relaxed standing | changes from baseline and after 6 weeks of intervention
  recorded in degree
Knee rotation angle in relaxed standing | changes from baseline and after 6 weeks of intervention
  recorded in degree

CONTACTS AND LOCATIONS:
Overall Officials: be945a7ts@gmail.com Chen, PhD, Study Director — National Yang Ming Chiao Tung University
Locations (1):
- National Yng Ming University, Taipei, 北投區, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis IS, Powers CM. Patellofemoral pain syndrome: proximal, distal, and local factors, an international retreat, April 30-May 2, 2009, Fells Point, Baltimore, MD. J Orthop Sports Phys Ther. 2010 Mar;40(3):A1-16. doi: 10.2519/jospt.2010.0302. No abstract available. PMID 20195028